CLINICAL TRIAL: NCT03689114
Title: Efficacy and Tolerability of Low vs. Standard Daily Doses of Antiepileptic Drugs in Newly Diagnosed, Previously Untreated Epilepsy (STANDLOW). A Multicenter, Randomized, Single-blind, Parallel-group Trial
Brief Title: Low vs. Standard Daily Doses of Antiepileptic Drugs in Newly Diagnosed, Previously Untreated Epilepsy(STANDLOW)
Acronym: STANDLOW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other); Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STANDLOW
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Epilepsies, Partial
Keywords: epilepsy; antiepileptic drugs; low dose; standard dose; new diagnosis
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Carbamazepine; Levetiracetam; Valproic Acid; Zonisamide; Oxcarbazepine; Topiramate; Lamotrigine; Gabapentin

STUDY DESIGN:
Intervention Model Description: This is a multicenter randomized pragmatic parallel-group single-blind non-inferiority trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental): Dosage is in mg: low dose carbamazepine, 300 ; low dose levetiracetam, 500; low dose valproate, 300; low dose zonisamide, 150; low dose oxcarbazepine, 600; low dose topiramate, 100; low dose lamotrigine, 100; low dose gabapentin, 450. Study drugs are in form of tablets for daily administration. Study drug administration duration is 12 months. The choice of the drug is left to the caring physician's discretion but it must be limited to the AEDs marketed for monotherapy use. All the study drugs will be used according to the respective SPCs, which will be sent by the promoter to all the study investigators.
  Interventions: Drug: Low dose carbamazepine; Drug: Low dose levetiracetam; Drug: Low dose valproate; Drug: Low dose zonisamide; Drug: Low dose oxcarbazepine; Drug: Low dose topiramate; Drug: Low dose lamotrigine; Drug: Low dose gabapentin
- Standard dose (Active Comparator): Dosage is in mg: standard dose carbamazepine 600; standard dose levetiracetam 1000; standard dose valproate, 600; standard dose zonisamide 300; standard dose oxcarbazepine 1200; standard dose topiramate, 200; standard dose lamotrigine, 200; standard dose gabapentin 900. Study drugs are in form of tablets for daily administration. Study drug administration duration is 12 months. The choice of the drug is left to the caring physician's discretion but it must be limited to the AEDs marketed for monotherapy use. All the study drugs will be used according to the respective SPCs, which will be sent by the promoter to all the study investigators.
  Interventions: Drug: Standard dose carbamazepine; Drug: Standard dose levetiracetam; Drug: Standard dose valproate; Drug: Standard dose zonisamide; Drug: Standard dose oxcarbazepine; Drug: Standard dose topiramate; Drug: Standard dose lamotrigine; Drug: Standard dose gabapentin

INTERVENTIONS:
Drug: Low dose carbamazepine — Carbamazepine, 300 mg/die
  Other Names: low carbamazepine
  Arms: Low dose
Drug: Standard dose carbamazepine — Carbamazepine 600 mg/die
  Other Names: Standard carbamazepine
  Arms: Standard dose
Drug: Low dose levetiracetam — Levetiracetam 500 mg/die
  Other Names: Low levetiracetam
  Arms: Low dose
Drug: Standard dose levetiracetam — Levetiracetam 1000 mg/die
  Other Names: Standard levetiracetam
  Arms: Standard dose
Drug: Low dose valproate — Valproate 300 mg/die
  Other Names: Low valproate
  Arms: Low dose
Drug: Standard dose valproate — Valproate 600 mg/die
  Other Names: Standard valproate
  Arms: Standard dose
Drug: Low dose zonisamide — Zonisamide 150 mg/die
  Other Names: Low zonisamide
  Arms: Low dose
Drug: Standard dose zonisamide — Zonisamide 300 mg/die
  Other Names: Standard zonisamide
  Arms: Standard dose
Drug: Low dose oxcarbazepine — Oxcarbazepine 600 mg/die
  Other Names: Low oxcarbazepine
  Arms: Low dose
Drug: Standard dose oxcarbazepine — Oxcarbazepine 1200 mg/die
  Other Names: Standard oxcarbazepine
  Arms: Standard dose
Drug: Low dose topiramate — Topiramate 100 mg/die
  Other Names: Low topiramate
  Arms: Low dose
Drug: Standard dose topiramate — Topiramate 200 mg/die
  Other Names: Standard topiramate
  Arms: Standard dose
Drug: Low dose lamotrigine — Lamotrigine 100 mg/die
  Other Names: Low lamotrigine
  Arms: Low dose
Drug: Standard dose lamotrigine — Lamotrigine 200 mg/die
  Other Names: Standard lamotrigine
  Arms: Standard dose
Drug: Low dose gabapentin — Gabapentin 450 mg/die
  Other Names: Low gabapentin
  Arms: Low dose
Drug: Standard dose gabapentin — Gabapentin 900 mg/die
  Other Names: Standard gabapentin
  Arms: Standard dose

SUMMARY:
There are no guidelines on the first maintenance daily dose of antiepileptic drugs (AEDs) in newly diagnosed, previously untreated epilepsy. Original trials and Cochrane reviews show that seizure remission can be achieved with differing daily doses. In clinical practice, the first maintenance dose varies significantly. In contrast, the risk of adverse treatment effects increases with dosage. There is thus the need to identify the lowest effective dose for treatment start. This background prompted us to undertake a randomized multicenter pragmatic non-inferiority trial comparing standard to low daily doses of AEDs to demonstrate that low doses are at least as effective as standard doses (as indicated by the national formulary) but are better tolerated and are associated with a better quality of life. If proven as effective as the standard dose, a low daily dose of AEDs is a benefit to the patient in terms of tolerability and safety and a source of savings for the National Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Newly diagnosed previously untreated epilepsy, defined according to the ILAE definition (Fisher et al, 2014);
3. Having experienced focal seizures, defined according to the ILAE criteria (Commission, 1981);
4. Able to understand and comply with the study requirements and release a written informed consent.

Exclusion Criteria:

A patient will be excluded if at least one of the following criteria will be met:

1. Age less than 18 years;
2. Having experienced primarily or secondarily generalized tonic and/or clonic seizures, or other (non-focal) seizure types;
3. Previous exposure to AEDs;
4. Requiring low or standard doses on account of individual needs;
5. Inability to understand the aims or modalities of the study;
6. Current pregnancy or planning to become pregnant during the study period (e.g. who are not post-menopausal, surgically sterile, or using inadequate birth control). A postmenopausal state is defined as no menses for 12 months without an alternative medical cause;
7. Previous treatment with an antiepileptic drug;
8. Men unable to practice contraception for the duration of the treatment.
9. Poor compliance with assigned treatments;
10. Refusal to release written informed consent;
11. The study investigators will receive the summary of product characteristics (SPC) available for each study drug. Patients cannot be enrolled in the study if the contraindications/warnings described in the SPC are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ettore Beghi, MD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- ASST Monza Ospedale San Gerardo, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abimbola S, Martiniuk AL, Hackett ML, Anderson CS. The influence of design and definition on the proportion of general epilepsy cohorts with remission and intractability. Neuroepidemiology. 2011;36(3):204-12. doi: 10.1159/000327497. Epub 2011 May 24. PMID 21606654
- [Background] Beghi E, Niero M, Roncolato M. Validity and reliability of the Italian version of the Quality-of-Life in Epilepsy Inventory (QOLIE-31). Seizure. 2005 Oct;14(7):452-8. doi: 10.1016/j.seizure.2005.07.008. Epub 2005 Aug 10. PMID 16098770
- [Background] Proposal for revised clinical and electroencephalographic classification of epileptic seizures. From the Commission on Classification and Terminology of the International League Against Epilepsy. Epilepsia. 1981 Aug;22(4):489-501. doi: 10.1111/j.1528-1157.1981.tb06159.x. No abstract available. PMID 6790275
- [Background] Fisher RS, Acevedo C, Arzimanoglou A, Bogacz A, Cross JH, Elger CE, Engel J Jr, Forsgren L, French JA, Glynn M, Hesdorffer DC, Lee BI, Mathern GW, Moshe SL, Perucca E, Scheffer IE, Tomson T, Watanabe M, Wiebe S. ILAE official report: a practical clinical definition of epilepsy. Epilepsia. 2014 Apr;55(4):475-82. doi: 10.1111/epi.12550. Epub 2014 Apr 14. PMID 24730690
- [Background] Gilliam F. Optimizing health outcomes in active epilepsy. Neurology. 2002 Apr 23;58(8 Suppl 5):S9-20. doi: 10.1212/wnl.58.8_suppl_5.s9. PMID 11971128
- [Background] Maguire M, Marson AG, Ramaratnam S. Epilepsy (partial). BMJ Clin Evid. 2010 Jun 28;2010:1214. PMID 21429248
- [Background] Perucca P, Jacoby A, Marson AG, Baker GA, Lane S, Benn EK, Thurman DJ, Hauser WA, Gilliam FG, Hesdorffer DC. Adverse antiepileptic drug effects in new-onset seizures: a case-control study. Neurology. 2011 Jan 18;76(3):273-9. doi: 10.1212/WNL.0b013e318207b073. PMID 21242496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The pre-planned sample size of 374 participants was not reached due to COVID-19 pandemic and difficulties of each center in satisfying the inclusion criteria. The total number of enrolled and randomized patients was 58.
Period: Overall Study
Arm/Group | Low Dose | Standard Dose
Started | 29 | 29
Completed | 27 | 25
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Standard Dose | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.6 [32.0 to 72.7] | 55.5 [35.3 to 71.2] | 54.9 [32.2 to 71.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 14 | 17 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 29 | 29 | 58
Type of seizures [Count of Participants; unit: Participants] — Included were only focal seizures based on ILAE classification
  Participants
    aware | 10 | 4 | 14
    impaired awareness | 19 | 25 | 44
Seizure frequency [Count of Participants; unit: Participants]
  <2/month | 20 | 21 | 41
  2-5/month | 4 | 4 | 8
  6-10/month | 2 | 1 | 3
  >10/month | 3 | 2 | 5
  not specified | 0 | 1 | 1
Etiology [Count of Participants; unit: Participants]
  Structural | 5 | 10 | 15
  Unknown | 24 | 19 | 43
PSQ-18 [Median (Inter-Quartile Range); unit: units on a scale] — Patients Satisfaction Questionnaire 18 items (PSQ-18) measures various aspects related to satisfaction in disease management (general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctors, accessibility and convenience), each with a range from 1 to 5, where 1 indicates the least possible satisfaction, 5 the greatest.
  units on a scale
    General satisfaction | 5 [4 to 5] | 4 [4 to 5] | 4 [4 to 5]
    Technical quality | 4 [4 to 5] | 4 [4 to 5] | 4 [4 to 5]
    Interpersonal manner | 4 [4 to 5] | 4 [4 to 5] | 4 [4 to 5]
    Communication | 4 [4 to 5] | 5 [4 to 5] | 4.5 [4 to 5]
    Financial aspects | 4 [3 to 5] | 4 [4 to 5] | 4 [3 to 5]
    Time spent with doctors | 4 [3 to 4] | 4 [3 to 4] | 4 [3 to 4]
    Accessibility and convenience | 4 [4 to 5] | 4 [3 to 5] | 4 [3 to 5]
Qolie 31 [Median (Inter-Quartile Range); unit: units on a scale] — The Quality-of-Life in Epilepsy Inventory (QOLIE-31) measures the quality of life in patients with epilepsy (range 0-100, where 0 indicates the worst quality of life, 100 the best).
  units on a scale | 69 [50 to 80] | 60 [46 to 65] | 64 [48 to 74]
Time from first symptoms to diagnosis [Median (Inter-Quartile Range); unit: months] | 5.7 [0.4 to 28.0] | 3.2 [0.1 to 21.5] | 4.6 [0.1 to 21.5]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: The proportion of patients experiencing a treatment failure motivated by the need to change the assigned dose or the assigned drug for seizure relapse during the follow-up.
  All proportions are reported as percentages.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 29 | 29
Participants | 11 | 11

2. Secondary Outcome: Drug-related Adverse Events
Description: the proportion of patients experiencing a treatment failure motivated by intolerable drug-related adverse events during the follow-up;
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 29 | 29
Participants | 3 | 3

3. Secondary Outcome: PSQ-18, Italian Version
Description: The score of the seven Patients Satisfaction Questionnaire 18 items (PSQ-18) subscales (general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, accessibility and convenience) at the last visit; the score of each subscale ranges from 1 (worst) to 5 (best).
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 20 | 17
units on a scale
  General satisfaction | 4.5 [3 to 5] | 4 [3 to 4]
  Technical quality | 4 [3.5 to 5] | 4 [4 to 4]
  Interpersonal manner | 5 [4 to 5] | 4 [3 to 5]
  Communication | 5 [3.5 to 5] | 4 [4 to 5]
  Financial aspects | 4.5 [4 to 5] | 4 [4 to 5]
  Time spent with doctors | 4 [3.5 to 4] | 4 [3 to 4]
  Accessibility and convenience | 4 [3.5 to 5] | 4 [4 to 4]

4. Secondary Outcome: QoLIE-31, Italian Version
Description: QoLIE-31 measures the quality of life of patients with epilepsy (range 0-100, where 0 corresponds to the worst quality of life and 100 corresponds to the best), at the end of study visit.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 20 | 18
units on a scale | 68 [56.5 to 76.5] | 64.5 [55 to 78]

5. Secondary Outcome: Health Care Resources Utilization.
Description: The mean daily patient's cost of health care resources consumed for the management of epilepsy during the first 12 months of the study.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: euro
Arm/Group | Low Dose | Standard Dose
Number analyzed (Participants) | 29 | 29
euro | 252.46 [167.90 to 252.46] | 474.50 [338.92 to 677.86]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Low Dose: Dosage is in mg: low dose carbamazepine, 300; low dose levetiracetam, 500; low dose valproate, 300; low dose zonisamide, 150; low dose oxcarbazepine, 600; low dose topiramate, 100; low dose lamotrigine, 100; low dose gabapentin, 450; low dose lacosamide 100 mg. Study drugs are in form of tablets for daily administration. Study drug administration duration is 12 months. The choice of the drug is left to the caring physician's discretion but it must be limited to the AEDs marketed for monotherapy use. All the study drugs will be used according to the respective SPCs, which will be sent by the promoter to all the study investigators.
  The arm/group "low dose" includes all the interventions listed above which correspond to low dose of each antiepileptic monotherapy.
  All the results were grouped by arm/group. In the adverse events tables all the single drugs were specified in each arm/group.
  The aim of this study was to compare the low dose arm/group versus the standard dose arm/group independently from the specific intervention/drug prescribed by the neurologist. Randomization was done by dose and not by drug. The drug has been chosen by the treating physician.
- Standard Dose: Dosage is in mg: standard dose carbamazepine 600; standard dose levetiracetam 1000; standard dose valproate, 600; standard dose zonisamide 300; standard dose oxcarbazepine 1200; standard dose topiramate, 200; standard dose lamotrigine, 200; standard dose gabapentin 900; standard dose lacosamide 200 mg. Study drugs are in form of tablets for daily administration. Study drug administration duration is 12 months. The choice of the drug is left to the caring physician's discretion but it must be limited to the AEDs marketed for monotherapy use. All the study drugs will be used according to the respective SPCs, which will be sent by the promoter to all the study investigators.
  The arm/group "standard dose" includes all the interventions listed above which correspond to standard dose of each antiepileptic monotherapy.
  All the results were grouped by arm/group. In the adverse events tables all the single drugs were specified in each arm/group.
  The aim of this study was to compare the low dose arm/group versus the standard dose arm/group independently from the specific intervention/drug prescribed by the neurologist. Randomization was done by dose and not by drug. The drug has been chosen by the treating physician.
Arm/Group | Low Dose | Standard Dose
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/29
Other Adverse Events (participants affected / at risk) | 9/29 | 11/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=29) | Standard Dose (N=29)
HEART FAILURE (Cardiac disorders) | 1 | 0 — Participant treated with Levetiracetam 500 mg (low dose)
DYSARTHRIA (Nervous system disorders) | 1 | 0 — Participant treated with Levetiracetam 500 mg (low dose)
OTHER, SPECIFY (Cardiac disorders) | 1 | 0 — Participant treated with Levetiracetam 500 mg (low dose)
status epilepticus (Nervous system disorders) | 0 | 1 — Participant treated with Lacosamide 200 mg (standard dose)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=29) | Standard Dose (N=29)
IRRITABILITY (Psychiatric disorders) | 1 (1) | 2 (2) — One participant was treated with levetiracetam 500 mg (low dose); two participants were treated with levetiracetam 1000 mg (standard dose)
Fatigue (Nervous system disorders) | 2 (2) | 3 (3) — One participants was treated with levetiracetam 500 mg (low dose), one was treated with oxcarbazepine 600 mg (low dose); two participants were treated with levetiracetam 1000 mg (standard dose), one with carbamazepine 600 mg (standard dose)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) — One participant was treated with oxcarbazepine 600 mg (low dose), one with lacosamide 100 mg (low dose).
rash maculo-papular (Eye disorders) | 0 (0) | 2 (2) — One participant was treated with carbamazepine 600 mg (standard dose) and one with oxcarbazepine 1200 mg (standard dose)
Somnolence (Nervous system disorders) | 4 (4) | 4 (4) — 2 participants were treated with levetiracetam 500 mg, 1 with oxcarbazepine 600 mg and 1 with lamotrigine 100 mg (low dose); 2 participants were treated with oxcarbazepine 1200 mg, 1 with levetiracetam 1000 mg, 1 with lacosamide 200 mg (standard).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03689114/Prot_SAP_000.pdf